CLINICAL TRIAL: NCT06235996
Title: Effects of Musical Intervention on Patient Pain and Anxiety for Office-based Procedures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lake Erie College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Rebecca Steiner, Ph.D., Principal Investigator, Lake Erie College of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2024-01-13; First posted 2024-02-01 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Pain management
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Primary Purpose: Treatment Allocation: Randomized Interventional Model: Parallel Assignment Masking: Not applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music Intervention (Experimental): A patient is scheduled for an office-based procedure such as a nerve block, epidural steroid injection, etc. Music-of-choice during the office-based procedure intervention is assigned to this group. Music via external speakers played in the procedure room. To ensure acute pain and anxiety control, participants will receive standard analgesic treatment in the beginning of their scheduled interventional procedure. Such treatment includes injection and topical application of lidocaine to induce local anesthesia. Standard of care is applied.
  Interventions: Procedure: Office-based procedure indicated for chronic pain with music
- Control (Other): A patient is scheduled for an office-based procedure such as a nerve block, epidural steroid injection, etc. No music intervention is assigned to this group. No music at any time during the procedure. To ensure acute pain and anxiety control, participants will receive standard analgesic treatment in the beginning of their scheduled interventional procedure. Such treatment includes injection and topical application of lidocaine to induce local anesthesia. Standard of care is applied.
  Interventions: Procedure: Office-based procedure indicated for chronic pain without music

INTERVENTIONS:
Procedure: Office-based procedure indicated for chronic pain with music — Such procedure may include sacroiliac joint (SI) steroidal injections, SI radiofrequency ablations, peripheral nerve stimulator implantations, caudal and laminar epidural steroidal injections, lumbar medial branch blocks, lumbar medial branch nerve radiofrequency ablations, spinal cord implantation of electro stimulators.
  Arms: Music Intervention
Procedure: Office-based procedure indicated for chronic pain without music — Office-based procedure indicated for chronic pain without music
  Arms: Control

SUMMARY:
The purpose of this study is to determine if the use of musical intervention reduces patient anxiety and provides a less painful experience during office-based procedures in a pain management clinic setting.

DETAILED DESCRIPTION:
100 patients who are scheduled for interventional procedures will be randomly assigned to either a music intervention group or a no-music group. Such interventional procedures include sacroiliac joint (SI) steroidal injections, SI radiofrequency ablations, peripheral nerve stimulator implantations, caudal and laminar epidural steroidal injections, lumbar medial branch blocks, lumbar medial branch nerve radiofrequency ablations, spinal cord implantation of electro stimulators. These procedures are fluoroscopically guided. Each group will consist of 50 participants. Participants in the music intervention group will listen to their preferred genre of music during their procedure. The study participants in the music intervention group will listen to music via external speakers played in the procedure room. The music will not be loud enough to disrupt the physician's communication with the patient. The no-music group will receive the same treatment throughout the procedure; however, this group will not listen to music at any time during the procedure. To ensure acute pain and anxiety control, participants in both groups will receive standard analgesic treatment in the beginning of their scheduled interventional procedure. Such treatment includes injection and topical application of lidocaine to induce local anesthesia. The patients in both groups will complete a questionnaire that contains VAS and STAI scoring metrics to measure pain and anxiety levels, respectively. This questionnaire will be completed before and immediately after the procedure. Furthermore, we will use salivary cortisol as a non-subjective biomarker of psychological stress in study subjects not undergoing corticosteroid injections. The saliva samples from the study participants will be collected before and after their scheduled office-based procedures. Upon collection of saliva samples from the study participants, the samples will be picked up by the LabCorp, which then will perform salivary cortisol testing; the results will be reported to the study team.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled office-based procedure
* Informed consent is signed by a subject

Exclusion Criteria:

* Major hearing impairment
* Sensitivity to music

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS score | Immediately before and after an office-based procedure
  Visual Analogue Scale (VAS) score
STAI score | Immediately before and after an office-based procedure
  State-Trait Anxiety Inventory (STAI) score
Blood pressure | Immediately before and after an office-based procedure
  Systolic and diastolic blood pressure
Heart rate | Immediately before and after an office-based procedure
  Heart rate
Biochemical marker of stress | Immediately before and after an office-based procedure
  Salivary cortisol levels

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Patel, MD, Study Director — NeuSpine Institute, Florida
Locations (2):
- United States (2):
  - NeuSpine Institute, Wesley Chapel, Florida
  - NeuSpine Institute, Zephyrhills, Florida

IPD SHARING:
Plan to Share IPD: No